CLINICAL TRIAL: NCT02846922
Title: Catheter Ablation Versus Rate Control in Patients With Atrial Fibrillation and Heart Failure: A Multicenter Study
Brief Title: Catheter Ablation and Rate Control of Atrial Fibrillation in Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jin Geng, MD, Nanjing Medical University
Other Study IDs: 20160020
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Catheter Ablation; Rate Control; Heart Failure; Atrial Fibrillation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- catheter ablation group: atrial fibrillation patients with heart failure who received catheter ablation for rhythm control
- rate control group: atrial fibrillation patients with heart failure who received pharmacological approaches for rate control

SUMMARY:
To evaluate the efficacy of catheter ablation and rate control in heart failure patients with atrial fibrillation.

DETAILED DESCRIPTION:
All patients received either catheter ablation for rhythm control or rate control before enrollment, and the investigators do not assign specific interventions to the subjects during the study. So this study might be considered to be observational.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* documented atrial fibrillation
* New York Heart Association Ⅱ-Ⅳ or left ventricular ejection fraction <50%

Exclusion Criteria:

* heart failure that had a suspected reversible cause
* previous ablation
* any contraindication to catheter ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coexisted with heart failure and atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | up to 3 years
  composite of all-cause mortality, stroke and unplanned hospitalization due to cardiovascular reasons

SECONDARY OUTCOMES:
all-cause mortality | up to 3 years
stroke | up to 3 years
  stroke must be certified by CT scan
unplanned hospitalization due to cardiovascular reasons | up to 3 years
  Unplanned hospitalization will be present only if the patient is hospitalized unexpectedly because of persisting or increasing complaints of heart failure and ventricular arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Jin Geng, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Bingjian Wang, MD, Study Chair — Huai'an First People's Hospital
Locations (1):
- Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No